CLINICAL TRIAL: NCT02508909
Title: Videoscopic Ilioinguinal Lymphadenectomy for Groin Lymph Node Metastases From Melanoma
Brief Title: Videoscopic Ilioinguinal Lymphadenectomy for Melanoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIDEO SIIO trial, 2011/41
Record Dates: First submitted 2015-07-16; First posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Melanoma; Secondary Malignant Neoplasm of Lymph Node
Keywords: Videoassisted surgery
MeSH Terms: conditions — Melanoma; Lymphatic Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Videoscopic ilioinguinal lymphadenectomy for melanoma (Experimental): Melanoma groin lymph node metastasis.
  Interventions: Procedure: Videoscopic ilioinguinal dissection

INTERVENTIONS:
Procedure: Videoscopic ilioinguinal dissection — Inguinal dissection is performed after subcutaneous inflation via three ports. Iliac dissection is obtained through a pro-peritoneal access.
  Other Names: Videoscopic groin lymphadenectomy

SUMMARY:
Groin lymph node dissection for melanoma patients is burdened by high post-operative morbidity, mainly related to wound. This is a prospective pilot trial investigated feasibility and postoperative outcomes of videoscopic ilioinguinal lymphadenectomy in patients with inguinal lymph node melanoma metastases.

DETAILED DESCRIPTION:
Videoscopic ilioinguinal dissection is a two-stage procedure. Dissection is performed using an ultrasound dissector. The inguinal step is performed via three ports (one 3-5 cm above the apex of the femoral triangle, a second 5 cm medial to the adductors, and the third 5 cm lateral to the Sartorius muscle). After subcutaneous inflation, a formal inguinal lymph node (LN) dissection is performed, removing the contents of the femoral triangle, with incision and removal of the femoral fascia and proximal and distal ligation of the saphenous vein with vascular endostaplers and endoclips. The specimen is extracted using an endobag from the incision of SLNB, which is systematically removed, or through a small enlargement of the incision of the apex trocar for patients with clinically positive LNs. The iliac step starts with open insertion in the pro-peritoneal space of a Hasson trocar, followed by positioning of two additional trocars (5 and 10 mm respectively) just laterally of the umbilical pubic line. After creation of pneumo-pelvis, the iliac femoral vessels are identified, isolated and all the external iliac LNs removed. Afterwards, the obturator LNs are dissected off the obturator nerve. LNs are retrieved with an endobag or directly through the 10mm trocar after insertion of protective endotrocar. Two drains are positioned at the end of procedure in the obturator fossa and in the inguinal space, respectively. Intra-operative and early post-operative outcome (lenght of stay, complications, number of LNs) is recorded. Follow-up consists in detection of any recurrence, measurement of lymphedema of the leg and evaluation of quality of life

ELIGIBILITY:
Inclusion Criteria:

Melanoma patients without distant metastasis and either positive SLNB or clinically positive inguinal lymph nodes

Exclusion Criteria:

American Society of Anaesthesiologists (ASA) classification III-IV Severe chronic obstructive pulmonary disease (COPD) and other restrictive lung disease, Severe ischemic heart disease and chronic heart failure Previous cerebral abnormalities (aneurysm/arteriovenous malformations, ischemic/hemorrhagic stroke, primary or secondary tumors), History of deep vein thrombosis (DVT) Childbearing state Severe hip functional limitation Previous hip/knee arthroplasty. Previous surgery in the groin region (e.g., hernia repair, great saphenous vein surgery, iliac-femoral bypass) was considered a contraindication only for the iliac stage of lymphadenectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Operative complications | 30 days
  Frequency, type and severity of operative complications according to the Clavien-Dindo classification. Grade I: no intervention required; Grade II: medical therapy resolved the complication; Grade III A: intervention without general anaesthesia; Grade III B: intervention under general anaesthesia.

SECONDARY OUTCOMES:
Leg lymphedema | Up to 12 months
  Lymphedema is measured pre-operatively at 3, 6 and 12 months after surgery. Number of patients with lymphedema according to the definition of the percent change > or = 7% of the sum of circumferences of the lower limb.
Quality of life | Up to 12 months
  Quality of life was evaluated with European Organization Research and Treatment of Cancer (EORTC)-Quality of Life Questionnaire (QLQ-C30) administered pre-operatively and after 3-6 and 9-12 months after surgery.This questionnaire is made up of 30 items to be later summarized in 5 functional scales, 3 symptom scales, 6 single items and a global health status scale. All of the scores are standardized using linear transformation and converted onto a 0-100 scale. Thus, a higher score for a functional scale and the global health status scale mean a high level of functioning/quality of life. Conversely, a high score for a symptom scale/item means a worse quality of life due to the symptoms perceived.
Recurrence | Up to 12 months
  Patients were re-evaluated 1, 3, 6, 9 and 12 months after surgery and every 6 months thereafter. Whole body CT scan and inguinal ultrasonography were performed every six months. Local, in-transit, regional and distant recurrences were recorded.
  Number of patients with histology confirmed local recurrence
Number of excised lymph nodes | 30 days
  Information extracted from pathology report. Implications for quality assurance monitoring.

REFERENCES:
- [Background] Sommariva A, Pasquali S, Rossi CR. Video endoscopic inguinal lymphadenectomy for lymph node metastasis from solid tumors. Eur J Surg Oncol. 2015 Mar;41(3):274-81. doi: 10.1016/j.ejso.2014.10.064. Epub 2014 Dec 27. PMID 25583458
- [Background] Martin BM, Etra JW, Russell MC, Rizzo M, Kooby DA, Staley CA, Master VA, Delman KA. Oncologic outcomes of patients undergoing videoscopic inguinal lymphadenectomy for metastatic melanoma. J Am Coll Surg. 2014 Apr;218(4):620-6. doi: 10.1016/j.jamcollsurg.2013.12.016. Epub 2013 Dec 24. PMID 24560569